CLINICAL TRIAL: NCT03757884
Title: Improving Medical-Decision Through Cognition, Technology and Communication, Phase 2
Brief Title: Medical Decisions in the Hospital Setting- M-Safety
Acronym: M-Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vineet Chopra, Chief, Division of Hospital Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00145793
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Diagnostic Errors
Keywords: Diagnostic Errors; Hospital Medicine

STUDY DESIGN:
Intervention Model Description: Pre-posttest study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Pod (Experimental): Mindfulness breathing, privacy screen, noise cancelling headphones, diagnostic checklist, diagnostic support on-line application
  Interventions: Behavioral: Mindfulness breathing exercise; Behavioral: Diagnostic Checklist; Behavioral: Noise cancelling headphones; Behavioral: Privacy tablescreen; Behavioral: Diagnostic assistance application

INTERVENTIONS:
Behavioral: Mindfulness breathing exercise — Spire monitor instructed mindfulness breathing
Behavioral: Diagnostic Checklist — Checklist reminder for diagnosis
Behavioral: Noise cancelling headphones — Noise cancelling headphones
Behavioral: Privacy tablescreen — Privacy Tablescreen
Behavioral: Diagnostic assistance application — Diagnostic assistance application

SUMMARY:
This project will introduce and evaluate an intervention designed to improve diagnostic decision making. The intervention will attempt to increase clinician mindfulness and reduce environmental distractions to promote focused thinking. A meta-cognitive intervention using a structured checklist will be evaluated to identify improvement in diagnostic and therapeutic decision-making and examine the role of mindfulness and architectural design in enhancing patient safety.

DETAILED DESCRIPTION:
This project will introduce and evaluate an intervention designed to improve diagnostic decision making. The intervention will attempt to increase clinician mindfulness and reduce environmental distractions to promote system 2 thinking. A meta-cognitive intervention using a structured checklist will be evaluated to identify improvement in diagnostic and therapeutic decision-making and examine the role of mindfulness and architectural design in enhancing patient safety.

This a pretest-posttest design study that will be conducted with hospitalist physicians working at Michigan Medicine and/or the VA Ann Arbor Healthcare System. The proposed intervention will provide the participants with tools to help promote mindfulness and focus to assist with the diagnostic process. To reduce distraction, headphones to block out surrounding noise and table screens to limit distractions will be offered. To assist with diagnosis, a diagnostic checklist and use of a IPad to use an online diagnosis application will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Medicine Physicians

Exclusion Criteria:

* Physicians other than Hopitalists

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Number of Patient Differential Diagnosis | 8 months
  Differential Diagnosis
Change in the Use of Diagnostic Checklist | 8 months
  Diagnostic Checklist

SECONDARY OUTCOMES:
Change in Mindfulness Behaviors Score | 8 months
  This 4 Question Survey Measures Characteristics of Mindfulness, Range- 1=Always, 6=Never
Change in Number of Patient Diagnostic Testing | 8 months
  Diagnostic Testing includes Laboratory and Imaging
Change in Time Participants are Measured as Calm | 8 months
  Time Measured in Minutes, Using the Spire Monitor
Change in Time Participants are Measured as Focused | 8 months
  Time Measured in Minutes, Using the Spire Monitor
Change in Time Participants are Measured as Tense | 8 months
  Time Measured in Minutes, Using the Spire Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Vineet I Chopra, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Ann Arbor VA Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Data security rules and regulations of the participating facilities (such as the University of Michigan and the Department of Veterans Affairs) will be followed. If data can be shared, all identifiers will be removed from the data. Data will be made available for research to those who request it once analyses has been conducted and findings have been published. Persons interested in using the data will need to submit a request in writing, stating their intended use.
Supporting Information: Study Protocol, ICF
Time Frame: Following completion of data analysis and manuscript publication
Access Criteria: Persons interested in using the data will need to submit a request in writing, stating their intended use. Requirements for sharing will include proof of IRB approval, acknowledgement in all publications of the funding source and of the study authors.

REFERENCES:
- [Background] Chopra V, Harrod M, Winter S, Forman J, Quinn M, Krein S, Fowler KE, Singh H, Saint S. Focused Ethnography of Diagnosis in Academic Medical Centers. J Hosp Med. 2018 Oct 1;13(10):668-672. doi: 10.12788/jhm.2966. Epub 2018 Apr 25. PMID 29694450
- See also: Patient Safety & Enhancement Program at the University of Michigan and the Ann Arbor VA Heathcare System — http://psep.med.umich.edu/

DOCUMENTS (1):
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03757884/ICF_000.pdf